CLINICAL TRIAL: NCT02310529
Title: Randomized Control Trial of an Interpersonal Psychotherapy for Maternal Depression
Brief Title: Interpersonal Psychotherapy for Maternal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PILL-IPT
Record Dates: First submitted 2014-11-15; First posted 2014-12-08 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Maternal Depression
Keywords: Maternal depression; Interpersonal Psycotherapy
MeSH Terms: interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interpersonal Psychotherapy (Experimental): Interpersonal Psychotherapy will be delivered to Intervention group. The intervention group will be further divided into 3 groups (8 depressed mothers in each group). IPT is 12-16 week treatment, contains a supportive element, an educational element, parenting element and an interpersonal relationship element. Its goals include helping mothers feel supportive, empowered and confident about their parenting abilities, which will directly influence in reducing their depressive symptoms as well as resolution of interpersonal conflicts. Groups will assist people who have become withdrawn, isolated and disconnected. Intervention will be delivered by trained clinical psychologists.
  Interventions: Behavioral: Interpersonal Psychotherapy
- Treatment as usual (No Intervention): Patients including in this group will be taking only treatment as usual (in Pakistan it means that participants attending in outpatients' clinic at regular intervals and may or may not be taking prescribed medication).

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy — Interpersonal Psychotherapy will be delivered to Intervention group. The intervention group will be further divided into 3 groups (8 depressed mothers in each group).IPT is 12-16 week treatment, contains a supportive element, an educational element, parenting element and an interpersonal relationship element. Its goals include helping mothers feel supportive, empowered and confident about their parenting abilities, which will directly influence in reducing their depressive symptoms as well as resolution of interpersonal conflicts. Groups will assist people who have become withdrawn, isolated and disconnected.
  Intervention will be delivered by trained clinical psychologists.
  Other Names: IPT
  Arms: Interpersonal Psychotherapy

SUMMARY:
Depression related to pregnancy frequently presents postpartum depression, which has deteriorating and lasting negative effects, not only on infant and child well being but also on mother's and father's mental health (Nancy K et al 2009). It is therefore important to introduce interventions aiming to improve mental health of mothers that could minimize the risk of diseases, and have positive effect child's on physical and psychological developmental wellbeing.

Therefore, this project has been designed to assess the effectiveness of Interpersonal Psychotherapy for Postnatal Depression in Pakistan.

DETAILED DESCRIPTION:
Prevalence of depression in the postnatal period is 10% to 17 % in western world ( O 'Hara and Swain 1996; Josseffson et al 2001; Yoshida et al 2001) and 23% to 36% in the developing world (Rahman et al 2003; Patel et al 2002; Husain et al 2006).

In developed countries, studies indicate that maternal depression is associated with long-term emotional, cognitive and behavioral problem in children. There is evidence of link between maternal psychopathology to physical health of child. Research evidence also indicates that long-term negative impact of postnatal depression is on the mother's mental health, on infant's development and on the marital relationship (Reay, Fisher, Robertson, Adams and Owen 2005).

because of high prevalence of maternal depression in low income countries like Pakistan, the present study is designed to test the effectiveness of Interpersonal Psychotherapy for women with maternal depression. The participants will be recruited from Civil hospital Karachi and also from three different communities. total 50 participants will be recruited and randomized to 2 groups: either intervention or TAU group. Assessment will be done on baseline, after completion of intervention and 3 months after completion of intervention. Assessment will include Edinburg Postnatal depression scale, Patient Health Questionnaire-9, Generalized Anxiety Disorder-7 and Rosenberg Self Esteem scale. Participants in intervention group will receive 12 sessions of Interpersonal Psychotherapy (IPT)

ELIGIBILITY:
Inclusion Criteria:

* Mothers age 18 years and above older with child below 3 years of age
* Meet the criteria for mild to moderate depressive symptoms on (EPDS (cut off score above 10) and
* Were resident of trial catchment area were included in the study.

Exclusion Criteria:

* Mothers who were suffering from severe depression, with diagnosed learning or physical disability or
* Any major psychiatric illness other than maternal depression, with Alcohol and substance dependent or
* Actively suicidal were excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Edinberg Postnatal Depression Scale (EPDS) To test the feasibility and acceptability of interpersonal psychotherapy in women suffering from postnatal depression. | 3 months
  EPDS will be used to assess depression

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 3 and 6 Months
  PHQ-9 will be used to assess severity of depression
Generalized Anxiety Disorder-7 (GAD-7) | 3 and 6 Months
  GAD-7 will be used to assess severity of anxiety
Rosenberg Self Esteem Scale (RSES) | 3 and 6 Months
  This scale will ne used to assess self esteem

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nusrat Husain, Study Director — PILL
Locations (4):
- Pakistan (4):
  - Civil hospital Karachi, Karachi, Sindh
  - Bhitaiabad, Karachi, Sindh
  - Bilal Colony, Karachi, Sindh
  - Yousuf Goth, Karachi, Sindh

REFERENCES:
- See also: Organizational Website — http://pill.org.pk